CLINICAL TRIAL: NCT01118897
Title: Concurrent Chemo-radiation Using Tomotherapy Based IMRT in Locally Advanced Gallbladder and Pancreatic Cancers :A Phase II Study
Brief Title: Tomotherapy in Locally Advanced Gallbladder and Pancreatic Cancers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Reena Engineer, Professor, Tata Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 599
Record Dates: First submitted 2010-05-03; First posted 2010-05-07 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2010-05

CONDITIONS: Pancreatic Neoplasms Malignant; Malignant Neoplasm of Gall Bladder Non-resectable
Keywords: Gall bladder; Pancreatic cancers; Tomotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neoadjuvant chemoradiation (Experimental): All patients will receive concurrent chemoradiation. Chemotherapy will consist of Inj. Gemcitabine 300mg/mt2 weekly throughout the course of Radiotherapy. Radiotherapy will be delivered using Tomotherapy to a dose of 57Gy/25# over 5 weeks
  Interventions: Radiation: Tomotherapy

INTERVENTIONS:
Radiation: Tomotherapy — Radiotherapy 57-60 Gy in 25 fraction to PTV boost (SIBV - simultaneous integrated Boost volume) (2.3-2.4Gy/Fr)
  Concurrent chemotherapy Weekly concurrent CT schedule: Inj Gemcitabine 300 mg/m2 weekly during RT.
  Surgery: All patients will be evaluated for surgery in the joint clinic by surgeons and other treating physicians at 6-8 weeks post CT-RT. PET CT Scan will be used as the imaging modality. Patients suitable for R0 resection will be planned for surgery. Inoperable patients will be treated with palliative chemotherapy.

SUMMARY:
SUMMARY

PROJECT TITLE: Concurrent chemo-radiation using Tomotherapy based IMRT in locally advanced Gallbladder and Pancreatic cancers: A Phase II study

SPECIFIC OBJECTIVES:

Primary To assess the radiological response by dose escalated IMRT in locally advanced inoperable gallbladder and pancreatic cancers.

Secondary

1. To assess the resectability rate with microscopic negative margin (R0).
2. To assess the acute and late toxicities (Number of Participants with Adverse Events as a Measure of Safety and Tolerability)
3. To study the locoregional control in the patients undergoing R0 resection
4. To study overall survival

DESIGN: Phase II study

STUDY POPULATION: All patients of age >18 years years diagnosed with non metastatic locally advanced inoperable gall bladder and pancreatic cancer

STUDY SIZE: 60 patients

METHODOLOGY: Sixty cases will be screened and taken for study if eligible after taking the informed consent.

Patients will receive radiotherapy using Tomotherapy based IMRT with concurrent chemotherapy Gemcitabine weekly. The response will evaluated at 6 weeks post chemoradiation and if operable will undergo surgery, if still inoperable or metastatic will receive palliative chemotherapy.

PROJECT PERIOD:

Total project period : 3 years Recruitment, Data collection : 2 years Complete analysis of data : 1 year

STUDY SITE: Tata memorial centre

DETAILED DESCRIPTION:
In both gall bladder and pancreatic cancer surgery is the main stay of treatment, but majority of these tumors are inoperable by virtue of adjacent organ infiltration. In this study, inoperable gallbladder and pancreatic cancer patients will be treated with high precision radiotherapy using Tomotherapy delivering higher dose of radiation along with chemotherapy. It is expected that this high dose precise radiotherapy along with chemotherapy will lead to good symptom relief and make some of these tumors operable.

ELIGIBILITY:
Inclusion Criteria:

1. Inoperable locally advanced gall bladder and pancreatic cancer by virtue of vascular encasement of superior mesenteric artery (SMA), celiac artery, hepatic artery, portal vein (PV) or deep hilar invasion precluding R0 resection.
2. Biopsy proven adenocarcinoma
3. KPS >= 70
4. Age >18 years
5. Medically fit for chemotherapy
6. Normal hematological, renal and hepatic function (Serum Bilirubin<3mg/dl)
7. No prior history of treatment with radiation or chemotherapy.
8. Patient willing and reliable for follow-up.

Exclusion criteria

1. Any other malignancy in any site.
2. Expected survival < 3months.
3. Severe co-morbid conditions ( Severe cardiac disorder, severe bronchial asthma, severely compromised liver function, psychological disorder)
4. Malignant ascitis.
5. Distant metastases by clinical examination or by imaging/whole bodyPET scan.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-12; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To assess the feasibility of concurrent chemo-radiation with dose escalated IMRT in locally advanced inoperable gallbladder and pancreatic cancers | 3 Years
  Number of Patients with Grade III adverse Events as a Measure of Safety and Tolerability

SECONDARY OUTCOMES:
Response to CTRT | 3 months
  All patients will undergo PET CT scan for radiological evaluation of response at 6 weeks post CTRT
R0 resection rate | 6 weeks
  All patients will be jointly evaluated for surgery 6 weeks post chemoradiation
Locoregional control | 3 years
Overall survival | 3 years
  At the median follow up of 3 years the 5 year overall survival rate would be assesed

CONTACTS AND LOCATIONS:
Overall Officials: Reena Engineer, MD, Principal Investigator — Tata Memorial Centre
Locations (1):
- Tata Memorial Centre, Mumbai, Maharashtra, India